CLINICAL TRIAL: NCT00014248
Title: A Phase I Study And Pharmacokinetics Of Adenosine 5'- Triphosphate (ATP) When Administered By Intravenous Infusion On A Multiple Weekly Dose Schedule To Patients With Advanced Malignancies (Solid Tumors)
Brief Title: Adenosine Triphosphate in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Supportive Care
Other Study IDs: CDR0000068522; DMS-0005; ATP-DMS-0005; NCI-G01-1923
Record Dates: First submitted 2001-04-10; First posted 2003-07-30 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Cachexia; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; cachexia
MeSH Terms: conditions — Cachexia | interventions — Adenosine Triphosphate

INTERVENTIONS:
Drug: adenosine triphosphate
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Adenosine triphosphate may decrease weight loss and improve muscle strength in patients with advanced solid tumors.

PURPOSE: Phase I trial to study the effectiveness of adenosine triphosphate in controlling loss of weight and loss of muscle mass in patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the individualized maximum tolerated dose of adenosine triphosphate in patients with advanced solid tumors.
* Determine the safety of this regimen in these patients.
* Determine the pharmacokinetics of this regimen in these patients.
* Determine the effect of this regimen on quality of life of these patients.
* Determine the influence of this regimen on cancer cachexia in terms of weight change, percentage of body fat, voluntary muscle strength, and plasma markers in these patients.
* Determine the effect of this regimen on tumor burden in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive adenosine triphosphate (ATP) IV over 8 hours on day 0. Treatment repeats weekly for a total of 8 courses in the absence of disease progression or unacceptable toxicity.

Each patient receives escalating doses of ATP until the individual maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which the patient experiences at least grade 3 (at least grade 2 cardiac ischemia or arrhythmia) toxicity.

Weight is measured at baseline and at weeks 1-8, 10, and 13. Percentage of body fat and skeletal muscle strength is measured at baseline and at weeks 2, 4, 8, 10, and 13.

Quality of life is assessed at baseline and at weeks 2, 4, 8, 10, and 13.

Patients are followed at weeks 10 and 13.

PROJECTED ACCRUAL: A maximum of 13-24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced solid tumor that is not curable by conventional therapy
* Brain metastases allowed if adequately controlled with radiotherapy

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 12 weeks

Hematopoietic:

* WBC at least 3,500/mm^3
* Absolute neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* SGOT and SGPT no greater than 3 times normal
* Bilirubin no greater than 2.0 mg/dL

Renal:

* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance greater than 60 mL/min
* BUN no greater than 25 mg/dL

Cardiovascular:

* Adequate cardiovascular function
* No congestive heart failure (New York Heart Association class III or IV heart disease)
* No angina pectoris AND/OR
* No significant arrhythmia
* No myocardial infarction within the past 6 months
* No clinically significant ischemic cardiac disease currently under treatment
* No clinically significant conduction system disease in the absence of a pacemaker (e.g., sick sinus syndrome, or second or third degree atrioventricular block)

Pulmonary:

* Adequate pulmonary function
* No clinical evidence of acute chronic obstructive pulmonary disease
* FEV1 at least 50% predicted
* Arterial oxygen tension at least 90% by pulse oximetry and on breathing room air
* No asthma OR
* No evidence of more than 20% reversibility in FEV1 with albuterol therapy

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No history of severe adverse reaction to adenosine
* No uncontrolled medical illness
* No average daily pain scores of at least 5 on a simple Visual Analogue Self pain assessment (0-10) scale

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Other:

* At least 30 days since prior investigational therapy
* At least 14 days since prior long-term theophylline, dipyridamole, or dipyridamole/aspirin therapy
* No concurrent long-term theophylline, dipyridamole, or dipyridamole/aspirin therapy
* No concurrent maintenance anti-anginal drug therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-10; Primary Completion 2002-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lionel D. Lewis, MD, Study Chair — Norris Cotton Cancer Center
Locations (1):
- Norris Cotton Cancer Center, Lebanon, New Hampshire, United States